CLINICAL TRIAL: NCT05149742
Title: Impact of Severe to Profound Deafness on Cognitive Functions in Middle-aged Adults
Brief Title: Deafness and Cognition in Middle-aged Adults
Acronym: SURDICOG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210439
Record Dates: First submitted 2021-10-28; First posted 2021-12-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment in Middle-aged Adults
Keywords: Severe and profound hearing loss; mild cognitive impairment (MCI); middle aged adult; depression
MeSH Terms: conditions — Cognitive Dysfunction; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases: Patients with severe to profound hearing loss (Experimental): Patients aged between 45 to 64 years with severe to profound bilateral post-lingual sensorineural hearing loss with a maximum intelligibility of 70% (disyllabic words) in free-field silence with hearing aids at 60 dB SPL
  Interventions: Behavioral: Cognitive and audiometry evaluation
- Controls: 90 matched subjects with normal hearing (Active Comparator): Healthy controls aged between 45 to 64 years with normal hearing on pure-tone audiometry (as function of ISO 7029 reference)
  Interventions: Behavioral: Cognitive and audiometry evaluation

INTERVENTIONS:
Behavioral: Cognitive and audiometry evaluation — For both Patients and controls:
  * Cognitive functions evaluation
  * Tonal and vocal audiometry
  * Self questionnaires

SUMMARY:
A mild cognitive impairment was observed in 50% of cochlear implant candidates aged 65 years and over, compared to 5-19% in general population. No studies analysed cognition in patients younger than 65 years. The aim of our study was to compare cognitive function between patients with severe and profound hearing loss and patients with normal hearing in patients aged 45 to 64 years.

DETAILED DESCRIPTION:
This case-control study will include 180 middle aged adults (90 cases, 90 healthy controls) matched on sex, age, education level in order to find an association between severe and profound hearing loss and presence of mild cognitive impairment.

90 subjects with severe to profound hearing loss,, with a maximum speech intelligibility of 70% for Fournier's disyllabic words in silence with properly fitted hearing aids could be included. Cognition evaluated on a battery of 5 tests, depression and dependance will be compared to healthy controls with normal hearing on pure-tone audiometry (as function of ISO 7029 reference) The subjects (cases and controls) will be recruited in the ENT consultation from the Cochlear Implant Center (Unité fonctionnelle implants auditifs, Pitié-Salpêtrière Hospital, Head: Dr Isabelle Mosnier)

ELIGIBILITY:
Inclusion Criteria:

* Cases: Patients aged between 45 to 64 years with severe to profound bilateral post-lingual sensorineural hearing loss with a maximum intelligibility of 70% (disyllabic words) in free-field silence with hearing aids at 60 dB SPL, current in french
* Controls: normal hearing subjects matched on age, sex and education level

Exclusion Criteria:

* Associated disability that prevents the tests from being performed
* Past and current history of neurological and psychiatric disorders including meningitis
* Psychotropic drug treatment
* Vulnerable subject

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-05-24 (Estimated); Study Completion 2027-05-24 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Mini Mental State Examination to access cognitive impairment in patients with severe to profound hearing loss compare to subjects with normal hearing | 1 day
  test to assess cognitive impairment. Result of this test is expressed on 30 points and is analyzed in function of age, sex, education level depending on publicised norms.
Evaluation of Trail making tests (TMT) A et B to evaluate executive functions in patients with severe to profound hearing loss compare to subjects with normal hearing | 1 day
  Trail making tests (TMT) A et B: rapidity test to evaluate executive functions. Score is expressed correct displacement number (in A and B parts) divided by time and multiply by ten.
Evaluation of "Fluences verbales sémantique et phonémique" to evaluate linguistic skills in patients with severe to profound hearing loss compare to subjects with normal hearing | 1 day
  "Fluences verbales sémantique et phonémique": test to evaluate linguistic skills. Score correspond to the number of words cited in 60 minutes in a specific category.
Evaluation of 16-item Free and Cue Selective Recall Test (RLRI/16) to evaluate episodic memory in patients with severe to profound hearing loss compare to subjects with normal hearing | 1 day
  16-item Free and Cue Selective Recall Test (RLRI/16): test adapted in French from the Free and Cue Selective Reminding test (FCSRT) assessing episodic memory. After an encoding phase during which the subject reads and memorizes 16 words 4 by 4, the subject is asked to freely recall as many words as possible in 2 minutes, cues are then provided. The free and cue recall is repeated 3 times and then 20 minutes later (delayed recall). The score used in the study will be: sum of the immediate free recall of the first three trials (0 to 48) and score of the delayed free recall (0 to 16)
Evaluation of Digit Symbol Substitution Test to evaluate psychomotor speed and executive functions, executive functions in patients with severe to profound hearing loss compare to subjects with normal hearing | 1 day
  Digit Symbol Substitution Test (DSST) of the Weschsler Adult Intelligence Scale-IV (WAIS-IV): test assessing attention, psychomotor speed and executive functions, executive functions. This test presents a matrix of nine digit-symbol pairs on a sheet of paper. A list of 135 numbers is presented in random order. The subject must associate the symbol corresponding to the number as quickly as possible by following the matrix. The score used will be: number of correctly associated symbols in 90 seconds
Evaluation of Instrumental activities of daily living scale to evaluate the level of dependence of dependence of the subjects in patients with severe to profound hearing loss compare to subjects with normal hearing | 1 day
  Instrumental activities of daily living scale (IADL): evaluation of the level of dependence of dependence of the subjects [45] (addendum 2). Patients with MCI must remain independent. The existence of dependence contributes to the diagnosis of of dementia
Evaluation of Cognitive Complaint Questionnaire to evaluate Cognitive assessment in patients with severe to profound hearing loss compare to subjects with normal hearing | 1 day
  Assessment or monitoring to be instituted for a score of 3 or more, and/or one "yes" answer to question 5, and/or two "yes" answers to questions: A,4,5,7,8.

SECONDARY OUTCOMES:
Type of MCI | 1 day
  Evaluate the type of MCI (amnesic, dysexecutive, multidomain)
Impact of the severity of the hearing loss on presence and severity of cognitive disorders | 1 day
  Subjective evaluation of hearing noise based on Speech and spatial questionnary : Patients have to mark a scale, for example with a cross, at the right place between 0 and 10. A mark on the value 10 means that he is perfectly capable of doing or experiencing what is described in the corresponding question. A mark on the 0 indicates that he/she is hardly able to do or experience what is described.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Dr MOSNIER, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre de Recherche en Audiologie (CReA) - Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No
All data will be collected and analysed into the GH Pitié-Salpêtrière (AP-HP)